CLINICAL TRIAL: NCT01320345
Title: A Randomised Trial to Evaluate the Efficacy on Retinopathy and Safety of Fenofibrate in Adults With Type 1 Diabetes. A Multicentre Double-blind Placebo-controlled Study in Australia and Internationally.
Brief Title: The Fenofibrate And Microvascular Events in Type 1 Diabetes Eye.
Acronym: FAME 1 EYE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Juvenile Diabetes Research Foundation Australia (Unknown); Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAME0001; ACTRN12611000249954 (Registry Identifier: Australian New Zealand Clinical Trials Registry (ANZCTR))
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes Mellitus; Diabetic Retinopathy; Diabetic Nephropathies
Keywords: Diabetes Mellitus; Type 1 Diabetes Mellitus; Retinopathy; Diabetic Nephropathy; Fenofibrate
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Retinopathy; Diabetic Nephropathies; Diabetes Mellitus; Retinal Diseases | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fenofibrate (Experimental): 145 mg tablet of fenofibrate administered daily for 36 months.
  Interventions: Drug: Fenofibrate
- Placebo (Placebo Comparator): Inert lactose tablet (otherwise matching active) administered daily for 36 months.
  Interventions: Drug: Inert lactose placebo

INTERVENTIONS:
Drug: Fenofibrate — 145 mg tablet of fenofibrate administered once daily for 36 months.
  Arms: Fenofibrate
Drug: Inert lactose placebo — Insert lactose tablet matching active tablet administered once daily for 36 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the potential benefits of 145 mg of daily fenofibrate in adults with type 1 diabetes mellitus and pre-existing non-proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
Diabetes is the most common cause of adult onset blindness. Irreversible vision loss is a most feared complication of diabetes. Fenofibrate is a blood fat lowering drug available in Australia and has been shown to reduce eye damage in people with Type 2 diabetes by 35-40%, and to prevent eye damage in Type 1 diabetic animal models. This study will evaluate the potential benefits of oral Fenofibrate 145mg once daily for average 36 months in 450 adults with Type 1 diabetes mellitus who are at high risk of eye damage.

ELIGIBILITY:
Inclusion criteria (for the main study):

1. Men or non-pregnant women (on acceptable contraception) with T1D* according to standard criteria:

   * T1D defined as either (1) T1D diagnosed below 40 years of age and insulin therapy commencing within one year of T1D diagnosis, or (2) T1D diagnosed before, at or after 40 years of age along with: i) Documented history of ketoacidosis, and/or ii) Documented history of very low or undetectable C-peptide (fasting <200 nmol/L or 0.2 pmol/L), and/or iii) Documented history of T1D related autoantibody/ies (anti-Glutamic acid decarboxylase, anti-A2, anti-ZnT8).
2. Age 18 years or over;
3. Estimated glomerular filtration rate (eGFR) must exceed 30 ml/min/1.73m2;
4. Must have at least one eligible eye with non-proliferative retinopathy (ETDRS score 35-53 inclusive) confirmed by current retinal photography within the last 3 months (irrespective of prior laser therapy). Note: Any eye having undergone prior pan-retinal laser therapy is not eligible, but prior focal, macular or grid laser does not exclude that eye from eligibility.;
5. All types of insulin therapy, with no restriction by level of HbA1c;
6. Willing and able to comply with all study requirements, including treatment, assessment and clinic visit attendances;
7. Able to personally read and understand the Participant Information and Consent Form and provide written, signed and dated informed consent to participate in the study.

Eligibility criteria for the reference group is limited to age and gender matched individuals who do not have T1D.

Exclusion criteria:

1. Definite indication for or contraindications to fibrate treatment (Other lipid drugs [e.g. statins, ezetimibe, fish oils] are allowed.);
2. Need for bilateral intra-ocular treatment or laser photocoagulation therapy within the next 3 months (this exclusion only applies to retinal laser photocoagulation treatment to the posterior pole i.e. laser correction of corneas for short-sightedness is NOT an exclusion criterion);
3. Prior bilateral pan-retinal photocoagulation (PRP) treatment for diabetic retinopathy;
4. Prior bilateral intra-ocular injection(s) within the last 6 months;
5. Bilateral cataract surgery within the last 6 months;
6. Planned bilateral cataract surgery within the next 12 months;
7. History of any other non-diabetic eye disease that is or is likely to affect bilateral vision;
8. History of photosensitive skin rash or myositis;
9. Abnormal thyroid function (untreated);
10. Liver function tests exceeding 3x upper limit of normal (ULN);
11. Persistent elevated unexplained blood creatinine phosphokinase level above normal range;
12. Documented fasting triglycerides (TG) levels >6.5 mmol/L;
13. History of pancreatitis, deep vein thrombosis (DVT) or pulmonary embolism;
14. Use of investigational drugs in the prior 8 weeks;
15. Any unstable condition in last 3 months including active sepsis, diabetic ketoacidosis;
16. Myocardial infarction (MI), unstable angina, stroke or heart failure within last 6 months;
17. Diagnosed cancer with ongoing treatment or prognosis anticipated at <5 years;
18. Any obstacle to regular follow-up including scheduled clinic attendances;
19. Prior or planned organ transplantation (including islet cells) with subsequent continued immunosuppression therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of clinical significant retinopathy progression. | As reported throughout the study and/or annual eye assessment post-randomisation
  Comprising 2-step progression of ETDRS score (to at least moderately severe grade), clinically significant macular oedema, need for laser surgery, need for intraocular anti-VEGF or corticosteroid therapy or vitrectomy, adjudicated to be for diabetic retinopathy (DR)

SECONDARY OUTCOMES:
The individual components of the primary endpoint | At baseline, 12 m post-randomisation, 24 m post-randomisation and the end of study visit (which is on average 36 months post-randomisation).
  Clinically significant retinopathy progression, 2-step progression of ETDRS score
Occurrence of clinically significant macula oedema (CSME). | As reported throughout the study
  Occurrence of clinically significant macula oedema (CSME) per standard ophthalmological assessment or laser therapy.
Need for laser surgery for DR | As reported throughout the study
  Need for laser surgery for DR
Need for intraocular anti-VEGF or corticosteroid injection or vitrectomy | As reported throughout the study
  Need for intraocular anti-VEGF or corticosteroid injection or vitrectomy for DR
Visual acuity. | At baseline, 12 m post-randomisation, 24 m post-randomisation and the end of study visit (which is on average 36 months post-randomisation).
  Visual acuity using ETDRS/LogMar or Snellen Chart
Macular volume and thickness | At baseline, 12 m post-randomisation, 24 m post-randomisation and the end of study visit (which is on average 36 months post-randomisation).
  Macular volume and thickness by Optical Coherence Tomography (OCT)
Albuminuria. | At baseline, 12 m post-randomisation, 24 m post-randomisation, the end of study visit (which is on average 36 months post-randomisation) and wash-out visit.
  Albuminuria measured as urinary albumin:creatinine ratio.
Estimated glomerular filtration rate. | At study completion and washout visit
  Estimated glomerular filtration rate using Modification of Diet in Renal Disease (MDRD) formula.
Peripheral neuropathy status | At baseline, 12 m post-randomisation, 24 m post-randomisation and the end of study visit (which is on average 36 months post-randomisation).
  Peripheral neuropathy status assessed by temperature & vibration sensation and monofilament test.
Autonomic neuropathy. | At baseline, 12 m post-randomisation, 24 m post-randomisation and the end of study visit (which is on average 36 months post-randomisation).
  Autonomic neuropathy (QTc and R-R intervals) on annual ECGs.
Total cardiovascular events. | As reported throughout the study.
  Total cardiovascular events including myocardial infarction, stroke, sudden cardiac death, hospitalisation for acute coronary syndrome or any revascularisation events.
Frequency of foot ulcer and non-traumatic amputation. | As reported throughout the study
  Foot ulcer and/or non-traumatic amputation are reported by site during the study.

OTHER OUTCOMES:
Lipid and lipoprotein levels | At baseline and end of study
  Lipid and lipoprotein levels
Biomarkers and molecular markers | At baseline and end of study
  Markers of inflammation, glycation and oxidative stress, angiogenesis and adipocyte function, and molecular markers, as change from baseline with study treatment
Quality of Life questionnaire | At baseline, 12 m post-randomisation, 24 m post-randomisation and the end of study visit
  Quality of Life questionnaire completed by participants annually

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Keech, Professor, Principal Investigator — NHMRC Clinical Trials Centre, The University of Sydney; Alicia Jenkins, Professor, Principal Investigator — NHMRC Clinical Trials Centre, The University of Sydney
Locations (24):
- Australia (20):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Garvan Institute of Medical Research, Darlinghurst, New South Wales
  - Retina Associates - South West Retina, Liverpool, New South Wales
  - Hunter Diabetes Centre, Merewether, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Cairns Hospital, Cairns, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Southern Adelaide Diabetes and Endocrine Services, Oaklands Park, South Australia
  - University Hospital Geelong, Geelong, Victoria
  - Heidelberg Repatriation Hospital, Heidelberg, Victoria
  - Baker Heart and Diabetes Institute, Melbourne, Victoria
  - St Vincent's Hospital Melbourne, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- New Zealand (2):
  - Auckland Diabetes Centre, Auckland
  - Christchurch Hospital, Christchurch
- Belfast Health and Social Care Trust, Belfast, United Kingdom